CLINICAL TRIAL: NCT06066151
Title: A Single Arm, Open-label Study of the Efficacy of Minayo Iron-rich Yeast Drink With SOD on Female Nutritional Anemia, Skin Condition and Qi-blood Deficiency Syndrome
Brief Title: The Efficacy of Minayo Iron-rich Yeast Drink With SOD on Female Nutritional Anemia, Skin Condition and Qi-blood Deficiency Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Agile Groups Network Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-RD-09-MY-001
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Anemia; Skin Condition
Keywords: Minayo Iron-rich Yeast Drink; SOD; GSH
MeSH Terms: conditions — Anemia; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Minayo Yeast Drink Product (Experimental): Minayo Iron-rich Yeast Drink with SOD, 385 pieces, 25ml/piece, each piece contains 13mg of iron.
  Main ingredients: Water, erythritol, jujube juice concentrate, Wolfberry juice concentrate, ferrous gluconate, olive powder, SOD yeast powder, yeast extract (including glutathione), artichoke, etc.
  Interventions: Dietary Supplement: Minayo Yeast Drink Product

INTERVENTIONS:
Dietary Supplement: Minayo Yeast Drink Product — Participants need to drink one piece of the products each day, for 4 consecutive weeks.

SUMMARY:
The goal of this single arm, open-label study is to learn about the efficacy of Minayo Iron-rich Yeast Drink with SOD on females who are aged 18-35 and suffer nutritional Anemia, skin condition and Qi-blood deficiency syndrome. The main question it aims to answer is:

- whether the serum ferritin level in blood is improved after the intervention

14 qualified participants will be enrolled to drink the product "Minayo Iron-rich Yeast Drink with SOD" for four weeks, once a day. Four site visits will be made for each participant so that all relevant clinical data will be captured and recorded for data analysis and reporting.

Researchers will compare the final blood test result (hemoglobin concentration level, Glutathione (GSH), Superoxide Dismutase (SOD)) against the baseline to conclude whether the product will be effective in improving Anemia and skin conditions.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 to 35;
* Hemoglobin concentration level below 110g/L based on WHO diagnostic criteria for anemia;
* Agree not to take any drugs, supplements, or other dairy products during the trial;
* Agree not to take any other medications or supplements containing iron during the trial;
* Willing to refrain from participating in other interventional clinical studies during the trial period;
* Be able to fully understand the purpose, benefits and potential risks including side effects of the research;
* Willing to obey all test requirements and procedures;
* Informed consent signed.

Exclusion Criteria:

* Anemia caused by organic diseases;
* Subject who is in the treatment of gastrointestinal symptoms;
* Lactose intolerance;
* Subject who is currently presence of other organic diseases affecting intestinal function, such as history of gastrointestinal resection, colon or rectal cancer, inflammatory bowel disease, diabetes, hyperthyroidism or hypothyroidism, congenital megacolon, scleroderma, anorexia nervosa, etc.;
* Controlling diet, exercising, or taking medications to control weight or affect appetite in the last 3 months;
* Subject who has any of the following medical history or clinical findings that may affect the evaluation of the trial effect: significant gastrointestinal disorders, liver, kidney, endocrine, hematological, respiratory and cardiovascular diseases;
* Abuse alcohol or other drugs, supplement or OTC drugs currently or n the past may cause bowel dysfunction or can affect test result evaluation;
* Frequently use of medications that may affect gastrointestinal function or the immune system according to investigator's judgment;
* Take laxatives or other substances that promote digestion 2 weeks before the trail start;
* Subject who used drugs or supplements of iron agent 10 days before the beginning of the trial;
* Pregnant or lactating women or those planning to become pregnant during the trial;
* PI deems that subjects could not fully cooperate with trial arrangements.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females, aged 18 to 35
Enrollment: 11 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change of Serum Ferritin Level | baseline day, end of week 4
  The change of serum ferritin level in blood, ng/mL (12~135ng/mL for healthy female, 27~375ng/mL for healthy male)

SECONDARY OUTCOMES:
Hemoglobin Concentration Level | baseline day, end of week 4
  The change of hemoglobin concentration level in blood, g/L (115-150g/L)
Superoxide Dismutase (SOD) Concentration Level | baseline day, end of week 4
  The change of Superoxide dismutase (SOD) concentration in blood, U/ml (1000~2000U/ml)
Glutathione (GSH) Concentration Level | baseline day, end of week 4
  The change of Glutathione (GSH) concentration level in blood, mg/L (280~380mg/L)
Skincare Measurement - Lines/Wrinkles | baseline day, end of week 4
  The changes of the lines/wrinkles on the face by Miravex Antera 3D imaging system

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Zhang, MD, Principal Investigator — Raison Biotech Co., Ltd.
Locations (1):
- Shanghai Raison CMA Lab, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No